CLINICAL TRIAL: NCT03097354
Title: Validation of the Assignment of Alcoholic Drinks to Predefined Drink Groups in the Composite International Diagnostic Interview (CIDI)
Brief Title: Assignment of Alcohol Drinks to CIDI Drink Categories
Acronym: AF-CIDI
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Sören Kuitunen-Paul, Research Assistant, Technische Universität Dresden
Other Study IDs: AF-CIDI
Record Dates: First submitted 2017-03-15; First posted 2017-03-31 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Drinking
Keywords: alcohol use; consumption measure; Composite International Diagnostic Interview (CIDI); internet survey; standardized assessment
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-students: Ad-hoc sample of German adults, not currently enrolled at a university, lifetime alcohol users, no intervention/observational survey study design
  Interventions: Other: no intervention/observational survey study design
- University students: Ad-hoc sample of German adults, currently enrolled at a university (most likely in Dresden, Germany), lifetime alcohol users, no intervention/observational survey study design
  Interventions: Other: no intervention/observational survey study design

INTERVENTIONS:
Other: no intervention/observational survey study design — no intervention/observational survey study design

SUMMARY:
Alcohol consumption is a prevalent behavior in Western societies, which may produce feelings of happiness and sociability, but also increases the risk of individual and societal detriments. A detailed knowledge about individual and region-specific alcohol consumption is crucial in many aspects of health systems, from general practitioner's diagnostic evaluation to decisions on health-care related fundings for prevention programs by legislative and executive councils.

The assessment of alcohol consumption often consists of questions like "What alcohol and in which amount did you drink lately?" which may be answered using a given list of prevalent alcoholic beverages. With this study, the investigators want to contribute to the understanding of psychological determinants in answering these questions. For example, it is not yet fully understood, to which extend and why certain beverages are assigned to one of several beverage groups. The investigators suspect that familiarity with specific beverages as well as product names may influence this assignment.

In this online survey, which is open to any German-speaking alcohol user no matter how often or how much alcohol one normally consumes, participants will be presented a list of common beverages (e.g. Cuba Libre, Prosecco, Weizen) and asked to assign these beverages to one of several beverage groups (e.g. whiskey, beer, sparkling wine).

DETAILED DESCRIPTION:
The investigators expect that alcohol users will assign alcoholic drinks based on the product names, which might lead to erroneous assignments to predefined drink groups in certain occasions (e.g. "Bierlikör - beer liquor"). Furthermore, it is hypothesized that this tendency is smaller the more familiar a user is with the drink. Lastly, it is hypothesized that drinks with relatively low use prevalence in the general population, e.g. sweet liquors and cocktails, and drinks that include alcohol mixed with non-alcoholic beverages (e.g. "Radler", a beer-lemonade mix), are more often subject to non-concordant assignment across participants compared to highly-prevalent drinks (e.g. "Pilsner").

Thus, the investigators expect alcohol users to:

1. assign >90% of the presented beverages correctly,
2. differ from the expert assignments especially in drinks they are not familiar with,
3. differ from the expert assignments especially in drinks with ambiguous names,
4. do not differ in their assignments based on their gender and age group.

ELIGIBILITY:
Inclusion Criteria:

* Lifetime-consumption of any of the 60 presented alcoholic beverages,
* Consumption of 12 or more alcoholic drinks past year,
* Ability to understand and accept the informed consent, to answer the presented questions and fill out all questionnaires

Exclusion Criteria:

* Multiple participation in this study
* not answering at least one presented questionnaire (60-beverages-questionnaire, assignment-questionnaire, AUDIT questionnaire, sociodemographic questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ad-hoc sample of German-speaking alcohol users, either currently studying at a university or not
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Beverage assignment | at the baseline survey
  Actual correctness of beverage assignment for each beverage (max. 60 beverages), either correct or incorrect

SECONDARY OUTCOMES:
Confidence | at the baseline survey
  Self-report of confidence in the specific beverage assignment (Answer categories: sure; medium; barely)
Familiarity | at the baseline survey
  Self-report of familiarity with the specific drink type (Answer categories: frequently consumed (>3 times); tried (1-3 times)

OTHER OUTCOMES:
Socio-demographics | at the baseline survey
  Gender, year of birth, German state/region, nationality, relationship status, education level, employment status,
Risk status for Alcohol Use Disorder | at the baseline survey
  Sum score of the 10-item AUDIT screening of the World Health Organization
Risky alcohol consumption | at the baseline survey
  Sum score of the first three AUDIT items, i.e. AUDIT-C score

CONTACTS AND LOCATIONS:
Overall Officials: Sören Kuitunen-Paul, Principal Investigator — Technische Universität Dresden
Locations (1):
- Institute of Clinical Psychology and Psychotherapy, Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kuitunen-Paul S, Kuitunen PT, Kadrić F, Lachenmeier DW, Čolić J, Leonhardt L, Scheffel C. Assignment of alcoholic beverages in the Munich Composite International Diagnostic Interview (M-CIDI): An online survey among German students and non-students. International Journal of Mental Health and Addiction. 2019;(ePub ahead of print). doi:10.1007/s11469-019-00074-5